CLINICAL TRIAL: NCT00765037
Title: Post Market Study on the Efficacy of the Encore Reverse Shoulder Prosthesis in a Small Group of Subjects
Brief Title: Retrospective Encore Reverse Shoulder Prosthesis Study
Status: Completed | Type: Observational
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Jane M. Jacob Ph.D., DJO Surgical
Other Study IDs: PS - 902
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Rotator Cuff Deficiency; Glenohumeral Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Encore RSP: Subjects who need treatment for rotator cuff deficiency or glenohumeral arthritis, received the Encore Reverse Shoulder Prosthesis and are willing to participate in the study.
  Interventions: Device: Encore Reverse Shoulder Prosthesis

INTERVENTIONS:
Device: Encore Reverse Shoulder Prosthesis — rotator cuff deficiency and glenohumeral arthritis

SUMMARY:
The purpose of this study is to evaluate the survivorship and efficacy of the Encore Reverse Shoulder Prosthesis in a group of no more than 50 subjects for whom data collection has already begun.

ELIGIBILITY:
Inclusion Criteria:

* The RSP is indicated for use in patients with a grossly rotator cuff deficient shoulder joint with severe arthropathy or a previously failed joint replacement with a grossly rotator cuff deficient shoulder joint.
* The patient's joint must be anatomically and structurally suited to receive the selected implant(s), and a functional deltoid muscle is necessary to use the device.
* The glenoid baseplate is intended for Cementless application with the addition of screws for fixation. The humeral stem is intended for cemented use only.

Exclusion Criteria:

* Infection or sepsis
* Insufficient bone quality which may affect the stability of the implant, as determined by the physician
* Muscular, neurological, or vascular deficiencies, which compromise the affected extremity
* Alcoholism or other addictions
* Materials (metals, etc) sensitivity
* Loss of ligamentous structures
* High levels of physical activity
* Non-functional deltoid muscle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who meet the indications for use of the RSP device AND who meet the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Kioschos, M.D., Principal Investigator — Nashville Orthopedic Specialists
Locations (1):
- Nashville Orthopedic Specialists, Nashville, Tennessee, United States

REFERENCES:
- See also: Sponsor Company home page — http://www.djosurgical.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Encore RSP
Started | 19 (Original number of eligible subjects who signed a consent form.)
Completed | 13 (Subjects who came in for 1 year visit.)
Not Completed | 6
Not completed — Lost to Follow-up | 5
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Encore RSP
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 75 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Survivorship of the Encore Reverse Shoulder Prosthesis
Description: Number of subjects who completed all study visits through the 1 year visit.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Encore RSP
Number analyzed (Participants) | 13
participants | 13

ADVERSE EVENTS:
Time Frame: The first subject was treated in 2005 and the final subject came in for their final follow-up visit in 2008. The study ran for 3 years but adverse events were only collected on subjects from their day of surgery through their one year follow-up visit.
Arm/Group | Encore RSP
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 11/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Encore RSP (N=19)
Back and Bilateral knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis and bladder infection (Renal and urinary disorders) | 1 (1)
Forearm and Jaw fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased left shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Increased right knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased right shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Left knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Multiple contusions (Injury, poisoning and procedural complications) | 1 (1)
Nasal fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Parkinson's Disease (Nervous system disorders) | 1 (1)
Right humeral fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Right middle trigger finger pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Right radial nerve palsy (Nervous system disorders) | 1 (1)
Right shoulder instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Staph infection at IV site (Infections and infestations) | 1 (1)
left elbow and hand pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less